CLINICAL TRIAL: NCT04943653
Title: Phase I,II Study of First Line Intraperitoneal Paclitaxel With Systemic Capecitabine and Oxaliplatin Combination Therapy in Patients With Advanced Gastric Cancer With Peritoneal Metastasis
Brief Title: Intraperitoneal Paclitaxel With XELOX in Gastric Cancer With Peritoneal Metastasis
Acronym: IPXELOX
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul St. Mary's Hospital (Other)
Responsible Party: Principal Investigator, In-ho Kim, Associate proffessor, Seoul St. Mary's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KC20MISF0813
Record Dates: First submitted 2021-06-21; First posted 2021-06-29 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-07

CONDITIONS: Stomach Neoplasms; Paclitaxel; Peritoneal Metastases
Keywords: Oxaliplatin; Capecitabine; XELOX
MeSH Terms: conditions — Stomach Neoplasms | interventions — Paclitaxel; Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intraperitoneal paclitaxel + XELOX (Experimental): Intraperitoneal paclitaxel Day1, Day8 + *XELOX
  *XELOX ; Capecitabine 2000mg/m2/day(Day1-14) Oxaliplatin 100mg/m2 IV Day1 q 3 weeks
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: Paclitaxel — intraperitoneal paclitaxel
  20mg/BSA(Body Surface Area), 40mg/BSA, 60mg/BSA (phase I)
  recommended dose (phase II)
  Other Names: capecitabine; oxaliplatin

SUMMARY:
IPXELOX will investigate the safety, tolerability, and antitumor activity of intraperitoneal paclitaxel in combination with chemotherapy in patients with advanced gastric cancer with peritoneal metastasis.

Study hypotheses: Intraperitoneal paclitaxel administered to subjects at the recommended phase 2 dose will show manageable safety and tolerability and anti-tumor efficacy with systemic capecitabine and oxaliplatin in advanced gastric cancer with peritoneal metastasis.

ELIGIBILITY:
1. Inclusion Criteria:

   * ECOG(Eastern Cooperative Oncology Group) performance status 0 or 1
   * pathologically proven primary gastric adenocarcinoma
   * peritoneal metastasis confirmed by laparoscopy or diagnostic imaging
   * written informed consent
   * adequate function of important organs (within 14 days before registration)

   Absolute neutrophil count ≥1.5 x 10^9/L, Platelet >=100,000/mm3, Hemoglobin >=8.0g/dL, Total bilirubin <= ≤ 2.0mg/dl or ULN(Upper Limit of Normal) x 1.5, AST(aspartate aminotransferase) <=100IU/L(International Unit/Liter), ALT(alanine transaminase) <=100IU/L, Creatinine clearance ≥ 50mL/min (milliliter/minute),
2. Exclusion Criteria:

   * other active concomitant malignancies
   * HER2(human epidermal growth factor receptor 2) positive (Immunohistochemistry 3+ or 2+ with in situ hybridization positive)
   * no investigational anticancer therapy within 30 days prior to the first dose of study treatment
   * recent (within 6 months) acute coronary syndrome, severe heart failure or severe pulmonary disease
   * uncontrolled acute or chronic disease
   * uncontrolled infection or inflammation
   * uncontrolled psychiatric disorder or central neurologic disease
   * not fully recovered from previous surgery
   * prior anticancer therapy (chemotherapy, immunotherapy, radiation) within 6 months
   * intolerable to oral administration or a lack of physical integration of the upper gastrointestinal tract or with a malabsorption syndrome
   * fertile males and females who are unwilling to use effective contraceptive methods.
   * pregnancy, breast feeding or intention to become pregnant
   * interstitial pneumonia or pulmonary fibrosis
   * peripheral neuropathy with functional impairment
   * hypersensitivity to paclitaxel, oxaliplatin, capecitabine, fluoropyrimidine or Cremophor EL.
   * concomitant therapy with any substrate or inhibitor of Cytochrome P450 2C8 or 3A4
   * concomitant therapy with sorivudine or brivudine
   * Dihydropyrimidine dehydrogenase (DPD) deficiency.
   * current or recent (within the 7 days prior to enrollment) treatment of tegafur-gimeracil-oteracil potassium

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Estimated)
Dates: Start 2021-06-08 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
6-month progression free survival (6-month PFS) | 6 months after start of treatment
  PFS is the time from date of first dose until the date of objective disease progression or death

SECONDARY OUTCOMES:
1-year overall survival (1-year OS) | 1 year after start of treatment
  OS is the time from date of first dose until death due to any cause
Objective Response Rate (ORR) | 6 months after start of treatment
  Confirmed ORR per RECIST 1.1 is the percentage of patients with Complete Response or Partial Response that is subsequently confirmed.
Conversion surgery rate | 6 months after start of treatment
  rate of conversion surgery
Ascites response | 6 months after start of treatment
  negative conversion rate of peritoneal cytology

CONTACTS AND LOCATIONS:
Locations (1):
- Gastric cancer center, Seoul St. Mary's Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No